CLINICAL TRIAL: NCT04818736
Title: COVID Vaccine for Indirect Protection: A Cluster Randomized Controlled Trial in Hutterite Colonies
Brief Title: COVID-19 Vaccine For Indirect Protection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Vaccine roll out plans increased so timing was no longer feasible
Sponsor: McMaster University (Other)
Collaborators: University of Alberta (Other); University of Saskatchewan (Other); University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-RCT
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-02

CONDITIONS: Vaccine Preventable Disease
Keywords: vaccination; herd immunity; COVID-19
MeSH Terms: conditions — Vaccine-Preventable Diseases; COVID-19 | interventions — heterologous prime boost COVID-19 vaccination; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- COVID-19 (Experimental): mRNA-1273 vaccine
  Interventions: Biological: COVID-19 Vaccination
- Control (Experimental): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Biological: COVID-19 Vaccination — Dose 1: 0.5 mL at Day 0 Dose 2: 0.5 mL at Day 28
  Other Names: Moderna mRNA-1273 vaccine
  Arms: COVID-19
Other: Usual care — Participants can receive the COVID-19 whenever they are eligible according to local provincial guidelines.
  Arms: Control

SUMMARY:
The primary objective of this study is to test whether vaccinating adults ≥18 years in Hutterite colonies with mRNA-1273 (Moderna COVID-19) vaccine as compared to control (usual care) can prevent RT-PCR confirmed COVID-19 in non-vaccinated Hutterite members.

DETAILED DESCRIPTION:
Despite the efficacy that has been demonstrated in Phase III randomized controls trials of mRNA COVID-19 vaccines, a critical question that remains unanswered is whether mRNA vaccines lead to herd immunity. The rationale for conducting this study is to learn whether vaccinating adults with a COVID-19 vaccine will prevent COVID-19 infections in non-vaccinated community members. Hutterite communities are unique since they are isolated from towns and cities and also share a number of communal activities, such as eating meals and attending church. Because of their location and practices, the Hutterite colonies give an opportunity to see whether vaccinating some Hutterite members with the COVID vaccine provides protection to the whole group. If the study shows that immunizing some of the population reduces the level of COVID-19 infection for other members of the population, this may be very important in stopping the COVID-19 pandemic and future pandemics.

ELIGIBILITY:
Group A: Anyone other than the adults aged ≥18 years who are vaccinated

Inclusion Criteria:

* Individuals under the age of 18
* Individuals with a contraindication to study vaccines
* Those not willing to be vaccinated but consent to follow up

Exclusion Criteria:

- There are no exclusion criteria for this category of participants:

Group B: Adults aged 18 years or older, who will be vaccinated as part of the intervention.

Exclusion Criteria:

* Anaphylactic reaction to any component of the study vaccine or to a previous dose of the study vaccines
* Pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
RT-PCR confirmed COVID-19 among non-vaccinated Hutterite colony members | 12 week period starting after first dose
  RT-PCR confirmed from nasal swabs

SECONDARY OUTCOMES:
RT-PCR confirmed COVID-19 among all Hutterite colony members | 12 week period starting after first dose
  RT-PCR confirmed from nasal swabs
RT-PCR confirmed COVID-19 in high-risk participants | 12 week period starting after first dose
  RT-PCR confirmed from nasal swabs
COVID-19 antibody testing | Baseline and through study completion, estimated at 4 months
  Blood spot testing of COVID-19 antibodies
Acute respiratory illness | 12 week period starting after first dose
  Participant self-report
School or work-related absenteeism | 12 week period starting after first dose
  Participant self-report
Physician visits for respiratory illness | 12 week period starting after first dose
  Participant self-report
Signs and symptoms of lower respiratory infection and pneumonia | 12 week period starting after first dose
  Participant self-report
Intensive care admission | 12 week period starting after first dose
  Participant self-report
Mechanical ventilation | 12 week period starting after first dose
  Participant self-report
Death | 12 week period starting after first dose
  Participant self-report

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No